CLINICAL TRIAL: NCT04222374
Title: Uro-DNA Collection for Expanded Genome-Wide Association Study (GWAS) of Renal Cell Carcinoma (RCC) (Uro-DNA - GWAS)
Brief Title: Uro-DNA Collection for Expanded Genome-Wide Association Study (GWAS) of Renal Cell Carcinoma (RCC)
Acronym: Uro-DNA - GWAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/20
Record Dates: First submitted 2019-12-09; First posted 2020-01-10 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2019-12

CONDITIONS: Kidney Cancer
Keywords: Renal Cell Carcinoma; Expanded Genome-Wide Association
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intervention in the UroCCR sites — 1. Blood sampling of a 5ml tube per patient. (for eligible patients recruited in the study, after signing the consent)
  2. DNA extraction:
     * For the patients of Bordeaux University Hospital, 2 aliquots will be constituted:
     * 1 aliquot for Expanded GWAS, containing at least 2 μg of DNA,
     * 1 aliquot for the UroCCR biobank.
     * For patients from other UroCCR centers, only 1 aliquot will be constituted:
     * 1 aliquot for Expanded GWAS, containing at least 2 μg of DNA.
  3. Transmission of the extracted DNA samples to the Biological Resource Center (CRB) of Bordeaux.
Procedure: Intervention in the CRB of Bordeaux University Hospital — 1. Temporary storage of DNA samples for Expanded GWAS before shipping to the NCI. Storage of samples for the DNA biobank.
  2. Overall packing of GWAS samples for shipment to the NCI.
  3. Shipping to the NCI: Constitutive DNA samples must be sent to the NCI by May 1, 2020 for inclusion in the Expanded GWAS study.
Procedure: Intervention at the Methodology and Data Management Centre of Bordeaux University Hospital — Transfer of the data associated with the samples to the NCI.
Procedure: Subsequent intervention at the NCI (for information) — 1. Samples will be genotyped at the NCI Cancer Genomics Research Lab using the Illumina Global Screening Network.
  2. GWAS combined meta-analysis, based, among others, on the results from the UroCCR samples.

SUMMARY:
In the last decade, investigators from the Department of Cancer Epidemiology and Genetics (National Cancer Institute, USA) have conducted genome-wide association (GWAS) studies of renal cell carcinoma.

Dr. Mark PURDUE and Dr. Stephen CAHNOCK (Department of Epidemiology of Cancer and Genetics, NCI) propose to expand their genome-wide association study (Expanded GWAS) by genotyping approximately 10,000 additional cases of kidney cancer patients, in collaboration with US institutions, South-American and European.

This study describes the participation of the French Kidney Cancer Research Network (UroCCR) in the Expanded GWAS research, under the coordination of Professor BERNHARD (Bordeaux University Hospital).

DETAILED DESCRIPTION:
The aim of the Expanded GWAS study is to better understand the role of common genetic variants in susceptibility to renal cell carcinoma (RCC).

The participation of the French UroCCR network consists in completing the bio-collection of the UroCCR cohort by preserving constitutional DNA and to provide DNA samples to the US NCI team.

This will increase the number of samples for meta-analysis and contribute to better identify clear cell kidney cancer susceptibility loci.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18,
* Confirmed cases of renal cell carcinoma (any RCC histology) of European or African origin,
* Patients included in the UroCCR study,
* Free, informed, written and signed consent by the participant and the investigator (at the latest on the day of inclusion and before any investigation required by the research) for specific blood collection for the purpose of DNA extraction,
* Programmed or ongoing management for kidney tumor,
* Constitutional DNA available (whole blood) for selected cases,
* Affiliated person or beneficiary of a social security scheme.

Exclusion Criteria:

* Patients below 18,
* Refusal of consent or participation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with kidney cancer included in the UroCCR project and coming for a regular consultation visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Identification of new clear cell Renal Cell Carcinoma (ccRCC) risk loci | Inclusion Visit
  From the DNA sample collected at inclusion visit, and the derived Single Nucleotide Polymorphisms (SNPs) genotype data:
  Association between evaluated genetic variants (SNPs) and renal cell carcinoma will be statistically determined if the p-value is found to be close to or lower than the Genome-wide significance threshold (p <5*10-8).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Talence, France

IPD SHARING:
Plan to Share IPD: No